CLINICAL TRIAL: NCT06920914
Title: Potassium (K) Handling in Advanced Chronic Kidney Disease (K-HANDLE CKD)
Brief Title: Effects of Minimally vs. Ultra-Processed Diets on Potassium (K) Handling in CKD
Acronym: K-HANDLE CKD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: Pro00139586; RES0062629 (Other Grant/Funding Number: Canadian Institutes of Health Research)
Record Dates: First submitted 2024-12-10; First posted 2025-04-10 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Chronic Kidney Disease
Keywords: CKD; Chronic Kidney Disease; potassium; hyperkalemia; hyperkalaemia; minimally processed foods; ultra-processed foods; feeding trial
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hyperkalemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Low-potassium, ultra-processed diet (Experimental): Participants in this group will follow a diet consisting of ultra-processed foods with restricted potassium content.
  Interventions: Other: Low-potassium, ultra-processed diet
- Normal potassium-rich, minimally processed diet (Experimental): Participants in this group will follow a diet consisting of minimally processed foods with a normal potassium content.
  Interventions: Other: Normal potassium-rich, minimally processed diet
- Normal potassium-rich, ultra-processed diet (Experimental): Participants in this group will follow a diet consisting of ultra-processed foods with a normal potassium content.
  Interventions: Other: Normal potassium-rich, ultra-processed diet
- Low-potassium, minimally processed diet (Experimental): Participants in this group will follow a diet consisting of minimally processed foods with restricted potassium content.
  Interventions: Other: Low-potassium, minimally processed diet

INTERVENTIONS:
Other: Low-potassium, ultra-processed diet — A diet restricted in potassium, primarily composed of industrially processed foods such as packaged snacks and processed meals.
  Arms: Low-potassium, ultra-processed diet
Other: Low-potassium, minimally processed diet — A diet restricted in naturally occurring potassium, primarily composed of fresh fruits, vegetables, whole grains, and other minimally processed foods.
  Arms: Low-potassium, minimally processed diet
Other: Normal potassium-rich, minimally processed diet — A diet with normal potassium content, primarily composed of fresh fruits, vegetables, whole grains, and other minimally processed foods, rich in naturally occurring potassium, following a Mediterranean-style pattern.
  Arms: Normal potassium-rich, minimally processed diet
Other: Normal potassium-rich, ultra-processed diet — A diet with normal potassium content, primarily composed of industrially processed foods such as packaged snacks and processed meals
  Arms: Normal potassium-rich, ultra-processed diet

SUMMARY:
What is this study about?

This clinical trial is designed to learn how potassium from different types of food affects blood potassium levels and overall health in people with chronic kidney disease (CKD, stages 3B-5).

People with CKD are often advised to avoid potassium-rich foods, even though fresh fruits and vegetables are important for good health. However, potassium in processed foods (such as packaged snacks and ready-made meals) may be absorbed differently than potassium from fresh foods.

This study will compare minimally processed vs. ultra-processed foods to determine how different sources of potassium affect potassium levels and help create better dietary recommendations for people with CKD.

What are the study goals?

The study will answer:

* Does potassium from fresh foods (like fruits and vegetables) affect blood potassium differently than potassium from processed foods?
* How does dietary potassium impact potassium absorption and excretion in people with CKD?

Researchers will compare the effects of four diets to understand how low and normal-potassium rich diets from fresh vs. processed foods influence:

* Blood potassium levels
* Body composition (muscle, fat, and fluid balance)
* Vascular health

What will participants do?

Participants will follow four different 10-day diets over the course of the study. All food will be provided at no cost. These diets are:

* Minimally processed with low-potassium content
* Minimally processed with normal potassium content
* Ultra-processed with with low-potassium content
* Ultra-processed with normal potassium content

There will be 16-day breaks (washout period) between diets where participants return to their normal eating habits.

During the study, participants will:

* Pick up prepared meals from the research center approximately 3 times per week.
* Attend checkups for weight, blood pressure, and blood tests.
* Provide urine samples to track potassium levels.
* Wear a comfortable, cuff-free blood pressure monitor at home.
* Keep a study journal to track diet, medications, and symptoms.
* Complete questionnaires about diet satisfaction and health changes.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged ≥18 years living with stage 3B-5 CKD (estimated glomerular filtration rate ≥ 15 mL/min/1.73m2) on conservative kidney management (not on dialysis).
* Able and willing to follow a controlled feeding regimen, attend in-person visits, provide informed consent, and comply with study procedures.

Exclusion Criteria:

General

* Pregnant or lactating women.
* Transitioning transgender individuals.
* Individuals with strict dietary preferences (e.g., vegetarians, vegans) or allergies/intolerance that would preclude participation in the diet phases.

Kidney Function

* Foreseen start of renal replacement therapy within the next 6 months.
* Acute kidney injury in the past 3 months.
* 2-year Kidney Failure Risk Equation > 40%.
* Preemptive kidney transplant planned within the next 6 months.
* History of kidney transplant.
* Active glomerulonephritis. Comorbidities
* Acute myocardial infarction or stroke within the past 6 months.
* Active cancer.
* Ileostomy, short bowel syndrome or inflammatory bowel disease.
* Body mass index < 18.5 or ≥ 35.
* New York Heart Association Class III or IV congestive heart failure.
* History of ventricular arrhythmia.
* Major surgery within the past 3 months.
* Active autoimmune disease.
* Glycated hemoglobin > 10% within the past 3 months.
* Gastroparesis.
* Chronic nausea and vomiting.
* Intensive care unit admission within the past 3 months.
* Significant psychiatric disease.
* Uncontrolled blood pressure (above 160/100). Current Use of Medications/Supplements
* Immunosuppressives.
* Potassium binders.
* Lithium.
* Motility agents.
* More than 2 medications that inhibit renal potassium excretion (e.g., angiotensin-converting enzyme inhibitors, angiotensin II receptor blockers, mineralocorticoid receptor antagonists).
* Supplements known to influence potassium levels. Potassium-Related Conditions
* Potassium > 5.5 mmol/L in more than 3 episodes within the past year.
* Participants with genetic issues affecting potassium handling (e.g. Barter and Liddle syndrome) or other unique health conditions that could interfere with potassium handling.

Intervention-related Conditions

* Fluid volume status or hypertension being actively managed. Other Factors
* Documented non-adherence to medications or other therapeutic measures.
* Use of tube feeding or parenteral nutrition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2026-07-01 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Fasting Serum Potassium Levels (mmol/L) | Days 10, 36, 62, and 88.
  This measure assesses the concentration of potassium in participants' blood after fasting overnight. Normal potassium levels typically range from 3.5 to 5.0 mmol/L.

SECONDARY OUTCOMES:
Postprandial Whole-Blood Potassium Response (mmol/L) | 15, 30, 60, 90, 120, 150, 180 minutes post-meal at days 10, 36, 62, and 88.
  This measure examines changes in blood potassium levels after a standardized test meal. Blood samples are collected before the meal (baseline) and at regular intervals (15, 30, 60, 90, 120, 150, and 180 minutes) to calculate the area under the curve (AUC), which reflects the total potassium response over time.
Potassium Bioavailability | Days 7-9, 33-35, 59-61, 85-87.
  Potassium bioavailability is assessed by measuring the potassium content in 24-hour urine samples. This provides insights into how much potassium from the diet is absorbed and how much is excreted by the body.
Body Composition (kg) | Baseline and days 10, 36, 62, and 88.
  This measure estimates participants' fat mass and fat-free mass. Body composition is assessed using bioelectrical impedance analysis, which uses safe, low-level electrical currents to estimate tissue and fluid distribution. Results are reported in kilograms (kg).
Body water (L) | Baseline and days 10, 36, 62, and 88.
  This measure evaluates fluid status, i which plays a role in potassium handling. Body water is estimated using bioelectrical impedance analysis, which uses safe, low-level electrical currents to estimate tissue and fluid distribution. Results are reported in liters for total, extracellular, and intracellular water.
24h blood pressure (mmHg) | Days 8-10, 34-36, 60-62, and 86-88.
  Systolic and diastolic blood pressure will be monitored for 24h.
Dietary Satisfaction Questionnaire | Days 10, 36, 62, and 88.
  Self-administered questionnaire to provide feedback on the palatability, variety, and overall acceptability of the study-provided diets.

OTHER OUTCOMES:
Hyperkalemic Events | Enrollment (Screening), baseline, and days 10, 36, 62, and 88.
  The frequency and severity of hyperkalemic events (serum potassium ≥5.5 mmol/L) are monitored throughout the study to ensure participant safety.
  Hyperkalemia episodes are recorded as a count of occurrences for each dietary phase. Evaluated at screening, baseline and Day 10 of each 10-day dietary phase.
Potassium Content in Foods (mg) | Before enrollment and through study completion, an average of 3 years
  The potassium content of study-provided meals is measured to ensure accurate dietary potassium levels during each phase. Measured during the menu development phase and throughout the study.
Phosphorus Content in Foods (mg) | Before enrollment and through study completion, an average of 3 years
  The phosphorus content of study-provided meals is measured to ensure accurate dietary phosphorus levels during each phase.Measured during the menu development phase and throughout the study.
Sodium Content in Foods (mg) | Before enrollment and through study completion, an average of 3 years
  The sodium content of study-provided meals is measured to ensure accurate dietary sodium levels during each phase. Measured during the menu development phase and throughout the study.

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Richard, PhD, Principal Investigator — University of Alberta; Branko Braam, MD, PhD, Principal Investigator — University of Alberta

IPD SHARING:
Plan to Share IPD: No
We have not yet finalized a plan for sharing individual participant data. The decision will depend on several factors, including participant consent, ethical approval, and institutional policies regarding data privacy and security. Future data sharing may be considered upon additional ethical review and participant consent.

REFERENCES:
- [Background] Picard K, Barreto Silva MI, Mager D, Richard C. Dietary Potassium Intake and Risk of Chronic Kidney Disease Progression in Predialysis Patients with Chronic Kidney Disease: A Systematic Review. Adv Nutr. 2020 Jul 1;11(4):1002-1015. doi: 10.1093/advances/nmaa027. PMID 32191264
- [Background] Picard K, Mager DR, Senior PA, Richard C. Potassium-Based Sodium Substitutes Impact the Sodium and Potassium Content of Foods. J Ren Nutr. 2025 Jan;35(1):64-71. doi: 10.1053/j.jrn.2024.05.010. Epub 2024 Jun 6. PMID 38848804
- [Background] Picard K. Potassium Additives and Bioavailability: Are We Missing Something in Hyperkalemia Management? J Ren Nutr. 2019 Jul;29(4):350-353. doi: 10.1053/j.jrn.2018.10.003. Epub 2018 Dec 19. PMID 30579674
- [Background] Picard K, Picard C, Mager DR, Richard C. Potassium content of the American food supply and implications for the management of hyperkalemia in dialysis: An analysis of the Branded Product Database. Semin Dial. 2024 Jul-Aug;37(4):307-316. doi: 10.1111/sdi.13007. Epub 2021 Jul 29. PMID 34323307
- [Background] Picard K RD BSc, Senior PA MBBS PhD FRCP(E) FRCP, Wilmott A BSc, Jindal K MD FRCPC, Richard C RD PhD, Mager DR RD PhD. Comparison of diet quality tools to assess nutritional adequacy for adults living with kidney disease. Can J Diet Pract Res. 2022 Dec 1;83(4):180-185. doi: 10.3148/cjdpr-2022-009. Epub 2022 May 3. PMID 35503893
- [Background] Picard K, Senior PA, Adame Perez S, Jindal K, Richard C, Mager DR. Low Mediterranean Diet scores are associated with reduced kidney function and health related quality of life but not other markers of cardiovascular risk in adults with diabetes and chronic kidney disease. Nutr Metab Cardiovasc Dis. 2021 May 6;31(5):1445-1453. doi: 10.1016/j.numecd.2021.02.002. Epub 2021 Feb 11. PMID 33812736
- [Background] Picard K, Griffiths M, Mager DR, Richard C. Handouts for Low-Potassium Diets Disproportionately Restrict Fruits and Vegetables. J Ren Nutr. 2021 Mar;31(2):210-214. doi: 10.1053/j.jrn.2020.07.001. Epub 2020 Aug 20. PMID 32830022